CLINICAL TRIAL: NCT04955717
Title: The Diagnosis and Treatment of Chlamydia Trachomatis and Neisseria Gonorrhoeae in Pregnant Women to Prevent Adverse Neonatal Consequences.
Brief Title: Antenatal Chlamydia Trachomatis and Neisseria Gonorrhoeae Testing to Prevent Adverse Neonatal Consequences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Botswana Harvard AIDS Institute Partnership (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeffrey D Klausner, Clinical Professor, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HS-21-00245
Record Dates: First submitted 2021-06-29; First posted 2021-07-09 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Chlamydia Trachomatis Infection; Neonatal Infection; Preterm Birth; Gonorrhea
Keywords: chlamydia trachomatis; neisseria gonorrhoeae
MeSH Terms: conditions — Premature Birth; Gonorrhea

STUDY DESIGN:
Intervention Model Description: Clinic randomized trial evaluating the effectiveness of antenatal CT and NG screening and treatment compared to the standard of care (treatment based on signs and symptoms) on pregnancy and neonatal outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Testing and treatment (Experimental): Participants will receive CT and NG testing and treatment (if necessary) at their first antenatal care visit and a visit during their third trimester. Women will also receive support for partner notification. All women will receive postnatal testing and treatment. Those who test positive at the postnatal visit will be offered infant testing.
  Interventions: Other: Chlamydia trachomatis and Neisseria gonorrhoeae screening using the GeneXpert
- Standard of care (No Intervention): Participants will receive the standard of care for STI management, which is treatment based on signs and symptoms. Women will also receive support for partner notification. All women will receive postnatal testing and treatment. Those who test positive at the postnatal visit will be offered infant testing.

INTERVENTIONS:
Other: Chlamydia trachomatis and Neisseria gonorrhoeae screening using the GeneXpert — Chlamydia trachomatis and Neisseria gonorrhoeae testing using the GeneXpert
  Arms: Testing and treatment

SUMMARY:
To assess the effectiveness of Chlamydia trachomatis (CT) and Neisseria gonorrhoeae (NG) testing and treatment during pregnancy to reduce adverse pregnancy and birth outcomes compared to the standard of care (treatment based on symptoms and signs).

DETAILED DESCRIPTION:
In this study investigators are conducting a two-arm, cluster randomized trial to assess the effectiveness of Chlamydia trachomatis (CT) and Neisseria gonorrhoeae (NG) testing and treatment during pregnancy to reduce adverse pregnancy and birth outcomes compared to the standard of care (treatment based on symptoms and signs). Investigators will enroll 500 asymptomatic pregnant women in the testing and treatment clinics, and they will receive CT and NG testing and appropriate treatment at their first antenatal care visit and at a visit during their third trimester. An additional 250 asymptomatic pregnant women will be enrolled in the standard of care clinics, and they will receive syndromic management with additional support for partner notification. All participants will be tested for CT and NG at the first postnatal visit and those who test positive will be offered infant testing. Investigators will determine if antenatal testing and treatment reduces maternal infections at delivery, preterm birth, low birth weight, and neonatal CT/NG infection. This study will provide evidence to help evaluate the effects of testing on vertical transmission and clinically important pregnancy neonatal health outcomes, and to evaluate and understand biological correlates of transmission.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 15 years,
* Currently pregnant,
* Attending first ANC visit,
* 27 weeks gestation or less
* Not currently experiencing CT/NG-related symptoms (determined by validated screening tool),
* Not treated for CT/NG in the past 30 days,
* Willingness to provide self-collected specimens for CT/NG testing (for the STI-testing group, this will take place at their first ANC visit, at another visit in their third trimester, and at postnatal care. For the standard of care group, samples will only be collected at postnatal care),
* Willingness to return for a test of cure if CT/NG test is positive during antenatal care,
* Will reside in Gaborone through the time of delivery and 1st postnatal visit,
* Willingness to have neonates tested for CT/NG at their first postnatal visit,
* Mentally competent to understand the informed consent.

Exclusion Criteria:

* Not mentally competent to understand study procedures or give informed consent,
* Individuals < 15 years,
* Men,
* Women who are not pregnant,
* Pregnant women not attending their first antenatal visit,
* Pregnant women at >27 weeks gestation
* Pregnant women with current STI-related symptoms (will receive standard of care),
* Treated for an STI in the past 30 days.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- University of Southern California, Los Angeles, California, United States
- DHMT Clinics, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

REFERENCES:
- [Derived] Mussa A, Wynn A, Ryan R, Babalola CM, Hansman E, Simon S, Bame B, Moshashane N, Masole M, Wilson ML, Klausner JD, Morroni C. Effect of antenatal Chlamydia trachomatis and Neisseria gonorrhoeae screening on postdelivery prevalence and vertical transmission in Gaborone, Botswana: findings from an exploratory study. Sex Transm Infect. 2025 Mar 24;101(2):81-87. doi: 10.1136/sextrans-2023-055965. PMID 39366745
- [Derived] Wynn A, Mussa A, Ryan R, Hansman E, Simon S, Bame B, Moreri-Ntshabele B, Ramogola-Masire D, Klausner JD, Morroni C. Evaluating the diagnosis and treatment of Chlamydia trachomatis and Neisseria gonorrhoeae in pregnant women to prevent adverse neonatal consequences in Gaborone, Botswana: protocol for the Maduo study. BMC Infect Dis. 2022 Mar 7;22(1):229. doi: 10.1186/s12879-022-07093-z. PMID 35255814

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinic
Period: Overall Study
Arm/Group | Testing and Treatment | Standard of Care
Started | 251; 4 Clinic | 249; 3 Clinic
Completed | 220; 4 Clinic | 207; 3 Clinic
Not Completed | 31; 0 Clinic | 42; 0 Clinic

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testing and Treatment | Standard of Care | Total
Number analyzed (Participants) | 251 | 249 | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 13 | 25
  Between 18 and 65 years | 239 | 236 | 475
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 28 [16 to 42] | 28 [17 to 42] | 28 [16 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 249 | 500
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 251 | 249 | 500
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Botswana | 251 | 249 | 500

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Diagnosed With C. Trachomatis and N. Gonorrhoeae Infection at Post-delivery
Description: Results from GeneXpert PCR screening for Chlamydia trachomatis (CT) or Neisseria gonorrhoeae (NG) infection among postpartum women up 12 weeks after birth outcome. We compare the proportion with CT and/or NG in both study arms
Time Frame: This outcome was assessed at the first postnatal care visit up to 12 weeks after delivery.
Measure: Count of Participants; unit: Participants
Groups:
- Testing and Treatment: Participants in the intervention will receive CT and NG testing and treatment (if necessary) at their first antenatal care visit and a visit during their third trimester. Women will also receive support for partner notification. All participants will receive postnatal testing and treatment. Those who test positive at the postnatal visit will be offered infant testing.
  Chlamydia trachomatis and Neisseria gonorrhoeae screening using the GeneXpert: Chlamydia trachomatis and Neisseria gonorrhoeae testing using the GeneXpert
Arm/Group | Testing and Treatment | Standard of Care
Number analyzed (Participants) | 206 | 187
Participants | 2 | 23

2. Secondary Outcome: Number of Neonates Diagnosed With Chlamydia Trachomatis or Neisseria Gonorrhoeae Infection at Post-delivery.
Description: Infants of mothers who tested positive for Chlamydia trachomatis or Neisseria gonorrhoeae infection at the first postnatal care visit will be tested using the GeneXpert PCR. We will compare the number of infected neonates between two arms.
Time Frame: This outcome will be assessed at the first postnatal care visit up to 12 weeks after delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Testing and Treatment | Standard of Care
Number analyzed (Participants) | 208 | 187
Participants | 7 | 3

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 36 weeks.
Description: All adverse events are reported to the IRB and, if appropriate, to the Data and Safety Monitoring Board (DSMB), or other government agencies.
Arm/Group | Testing and Treatment | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/251 | 1/249
Serious Adverse Events (participants affected / at risk) | 16/251 | 15/249
Other Adverse Events (participants affected / at risk) | 0/251 | 0/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testing and Treatment (N=251) | Standard of Care (N=249)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 9 (9) — Defined as pregnancy loss before the 20th week of gestation wa identified through self-report by the participants, and through medical record abstraction.
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 6 (6) — Defined as fetal death at or after 20 weeks gestation and prior to delivery, was identified through self-report by the participants, and medical record abstraction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT04955717/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT04955717/SAP_001.pdf